CLINICAL TRIAL: NCT06925802
Title: Osteopathic Visceral Manipulation on Functional Constipation in Obese Adults: Randomized Controlled Clinical Trial
Brief Title: Osteopathic Visceral Manipulation on Functional Constipation in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assisstant professor, MTI University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB # 22 /3 / 2024-2025
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Constipation - Functional

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- osteopathic visceral manipulation (Experimental): Group A received osteopathic visceral manipulation with standard care
  Interventions: Other: visceral manipulation
- control (No Intervention): Group B received standard care only

INTERVENTIONS:
Other: visceral manipulation — The procedure begins with the patient lying in a comfortable supine position to ensure relaxation and access to the abdominal region. Gentle palpation is used to assess tissue mobility and identify any restrictions or tension points. The practitioner applies light, rhythmic pressure to the gastroduodenal junction to stimulate movement and improve coordination between the stomach and duodenum. Attention is then given to the sphincter of Oddi, where soft, sustained pressure is employed to facilitate the release of bile and pancreatic juices, aiding digestive processes. Moving to the duodenojejunal flexure, the therapist uses gentle stretching and mobilization techniques to alleviate any obstructions, promoting smoother passage of intestinal contents. Finally, the sigmoid colon is manipulated with circular and oscillatory pressures to enhance peristalsis and relieve constipation.
  Other Names: standard care only
  Arms: osteopathic visceral manipulation

SUMMARY:
Functional constipation in obese adults is a prevalent gastrointestinal issue characterized by infrequent bowel movements, difficulty during defecation, or a sensation of incomplete evacuation. Obesity is a significant risk factor for functional constipation due to several physiological and lifestyle-related factors. Excess body weight, particularly in the abdominal region, may exert pressure on the colon, leading to disrupted bowel function. Additionally, dietary habits common among obese individuals, such as low fiber intake and inadequate hydration, can worsen constipation. Sedentary lifestyles further contribute to reduced gastrointestinal motility. Addressing functional constipation in obese adults requires a multifaceted approach, including dietary modifications to increase fiber and fluid intake, regular physical activity, and, in some cases, medical interventions to alleviate symptoms and improve quality of life.

DETAILED DESCRIPTION:
Visceral manipulation is a gentle manual therapy that focuses on the internal organs, particularly those within the gastrointestinal tract, to enhance their function and alleviate symptoms associated with various disorders. Practitioners of visceral manipulation use their hands to apply specific, subtle forces to the affected areas, aiming to improve the mobility and motility of the organs. This technique is based on the premise that the body's organs are interconnected by fascia and ligaments, and any restriction or imbalance in these connections can lead to dysfunction and disease. By restoring the natural movement of these organs, visceral manipulation is believed to improve blood circulation, enhance digestive function, and reduce pain and discomfort associated with gastrointestinal disorders.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with functional constipation according to Rome IV criteria
* Body mass index (BMI) ≥ 30 kg/m²
* Ability to provide informed consent

Exclusion Criteria:

* patients with organic gastrointestinal diseases, Pregnancy or lactation
* Participation in another clinical trial within the last 30 days, Endocrine and metabolic disorders (eg, hypothyroidism, hypercalcemia, diabetes mellitus, diabetes insipidus)
* Neurologic and psychiatric disorders (spina bifida, cerebral palsy, anorexia nervosa, known autism spectrum disorders)
* Secondary constipation to drug consumption, History of abdominal surgery

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Stool consistency | at baseline and at three weeks
  Patients were asked to describe the consistency of their stools during the previous month, choosing between the terms "hard or very hard," "not too hard, not too soft (normal)," "soft or very soft," "mucous, with undigested food," and "liquid," they also had the opportunity to answer that the stools were "variable" in consistency. In addition, patients were asked to choose the BSS stool type that best represented their stools on a picture chart
Defecation Pain | at baseline and at three weeks
  Clearly explain to the patient the purpose of assessing their defecation pain using Arabic version of Visual Analogue Scale (VAS) form: A horizontal or vertical line, typically 10 centimeters in length, anchored by two descriptors at each end representing "no pain" and "worst possible pain."

SECONDARY OUTCOMES:
Defecation frequency | at baseline and at three weeks
  Utilize a standardized stool diary where participants record each defecation event, including the date
Dose of oral laxative | at baseline and at three weeks
  dose of oral laxative and time. Ensure the diary is easy to use to promote accurate self-reporting. Supplement diary entries with qualitative interviews to understand lifestyle, dietary habits, and stress levels, which may influence bowel movement

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No